CLINICAL TRIAL: NCT00818909
Title: Study to Evaluate the Physical Effect of SYSTANE QID in People That Have Moderate to Severe Dry Feeling Eyes
Brief Title: Systane Clinical Experience Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARES-3
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye; Systane; Moderate to severe dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane (Experimental): Systane ocular product
  Interventions: Other: Systane

INTERVENTIONS:
Other: Systane — Systane prescription

SUMMARY:
To evaluate the physical effect of SYSTANE QID in people that have moderate to severe dry eyes and to establish doctor confidence to prescribe Systane.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe dry feeling eyes

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
corneal and conjunctiva staining score | 4 weeks

SECONDARY OUTCOMES:
Tear film break up time | 4 weeks